CLINICAL TRIAL: NCT02045732
Title: A Phase 1b, Double-blinded, Placebo-controlled, Randomized Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Ascending Doses Of Pf-06342674 (rn168) In Subjects With Multiple Sclerosis (ms)
Brief Title: A Study To Evaluate The Safety And Tolerability Of PF-06342674 (RN168) In Subjects With Multiple Sclerosis (MS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study terminated on April 8, 2015 due to a corporate decision and not related to the safety or efficacy of the protocol.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B4351002
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MRI
MeSH Terms: conditions — Multiple Sclerosis | interventions — monoclonal antibody RN168

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Biological: PF-06342674 0.25 mg/kg; Biological: Placebo
- PF-06342674 1.5 mg/kg (Experimental)
  Interventions: Biological: Placebo; Biological: PF-06342674 1.5 mg/kg
- PF-06342674 6.0 mg/kg (q2 Weeks) (Experimental)
  Interventions: Biological: Placebo; Biological: PF-06342674 6.0 mg/kg
- PF-06342674 6.0 mg/kg (q1 Week) (Experimental)
  Interventions: Biological: Placebo; Biological: PF-06342674 6.0 mg/kg

INTERVENTIONS:
Biological: PF-06342674 0.25 mg/kg — Bi-Weekly Subcutaneous Injections X 6
  Arms: Cohort 1
Biological: Placebo — Bi-Weekly Subcutaneous Injections X 6
Biological: PF-06342674 1.5 mg/kg — Bi-Weekly Subcutaneous Injections X 6
  Arms: PF-06342674 1.5 mg/kg
Biological: PF-06342674 6.0 mg/kg — Bi-Weekly Subcutaneous Injections X 6
  Arms: PF-06342674 6.0 mg/kg (q1 Week); PF-06342674 6.0 mg/kg (q2 Weeks)

SUMMARY:
PF-06342674 (RN168), being developed for the treatment of multiple sclerosis (MS), is an antibody that binds to and inhibits the human interleukin-7 receptor, a component potentially involved in MS. PF-06342674 (RN168) is expected to play a role in slowing down the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-55 yrs.
* Confirmed diagnosis of Multiple Sclerosis (MS) according to the 2010 revision of the McDonald Criteria.
* Expanded Disability Status Scale (EDSS) between 0-5, inclusive.

Exclusion Criteria:

* Relapse episode of MS within 2 weeks of enrollment.
* Primary progressive MS without a relapsing component.
* Intolerant or unwilling to undergo MRI scanning. Treatment with disease modifying agents up to 6 weeks prior to enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Albany Advanced Imaging, Albany, New York
  - Fallon Wellness Pharmacy, Latham, New York
  - Northeast Eye Center, Latham, New York
  - The MS Center of Northeastern New York, Latham, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Radiology Associates (X-ray facility only), Oklahoma City, Oklahoma

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4351002&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20PF-06342674%20%28RN168%29%20In%20Subjects%20with%20Multiple%20Sclerosis%20%28MS%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a Phase 1b, randomized, multi-center, double-blind, sponsor-open, placebo controlled study to evaluate multiple ascending doses of PF-06342674 in participants with Multiple Sclerosis (MS). Up to 60 participants were planned to be enrolled. However, only 4 participants were randomized due to the early termination of the study.
Pre-assignment Details: Participants were screened within 45 days prior to the first administration of the study drug to confirm that they met the participant inclusion criteria for the study.
Groups:
- Placebo: Participants received placebo subcutaneously (SC) every other week during an 85-day treatment period.
- PF-06342674 0.25 mg/kg: Participants received PF-06342674 0.25 milligram (mg)/kilogram (kg) SC every other week during an 85-day treatment period.
Period: Overall Study
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Started | 1 | 3
Completed | 0 | 2
Not Completed | 1 | 1
Not completed — At the discretion of the investigator | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo SC every other week during an 85-day treatment period.
- PF-06342674 0.25 mg/kg: Participants received PF-06342674 0.25 mg/kg SC every other week during an 85-day treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06342674 0.25 mg/kg | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (0) | 45.3 (14.2) | 42.3 (13.1)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), and Withdrawals Due to AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study drug and up to Day 127/Early Termination that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline through Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
participants
  AEs | 0 | 3
  SAEs | 0 | 0
  Withdrawals Due to AEs | 0 | 0

2. Primary Outcome: Number of Treatment-Emergent AEs and SAEs by Severity
Description: AE severity was graded as mild, moderate, or severe. Mild AEs do not interfere with the participant's usual function. Moderate AEs interfere to some extent with the participant's usual function. Severe AEs interfere significantly with the participant's usual function.
Time Frame: Baseline through Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug.
Measure: Number; unit: adverse events
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
adverse events
  Mild | 0 | 7
  Moderate | 0 | 0
  Severe | 0 | 0

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality. Laboratory test parameters included hematology, liver function, renal function, electrolytes, hormones, clinical chemistry, and urinalysis (dipstick and microscopy). Abnormal laboratory findings included: lymphocytes (absolute) less than (<)0.8 x lower limit of normal (LLN); urine blood/hemoglobin (qualitative) more than or equal to (>=)1; urine nitrite >=1; urine leukocyte esterase >=1; urine red blood cell (RBC) >=20/high-power field (HPF).
Time Frame: Baseline through Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
participants | 0 | 3

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Categorical summarization criteria in vital signs included: supine systolic blood pressure (SBP) of <90 millimeters of mercury (mm Hg) or change in supine SBP of >=30 mm Hg; supine diastolic blood pressure (DBP) of <50 mm Hg or change in supine DBP of >=20 mm Hg; supine pulse rate of <40 or more than (>)120 beats per minute (bpm).
Time Frame: Baseline through Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
participants
  Supine SBP <90 mm Hg | 0 | 0
  Supine DBP <50 mm Hg | 0 | 0
  Increase in supine SBP >=30 mm Hg | 0 | 0
  Decrease in supine SBP >=30 mm Hg | 0 | 0
  Increase in supine DBP >=20 mm Hg | 0 | 0
  Decrease in supine DBP >=20 mm Hg | 0 | 0
  Supine pulse rate <40 bpm | 0 | 0
  Supine pulse rate >120 bpm | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: Criteria for potential clinical concern in ECG parameters: The maximum of the beginning of the Q wave to the end of the T wave corresponding to electrical systole (QT) interval corrected using the Fridericia formula (QTcF) >=450 milliseconds (msec), maximum QTcF interval change from baseline in range of 30 to <60 msec and >=60 msec.
Time Frame: Baseline through Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug. The QTcF interval of the participant in the placebo arm was in this range of 450 to <480 msec at Baseline. This participant experienced a decrease in QTcF of 30 to <60 msec on Day 30, which then returned to baseline levels on Day 57.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
participants
  QTcF Interval 450-<480 msec | 1 | 0
  QTcF Interval >=480 msec | 0 | 0
  QTcF Interval 30-<60 msec Increase From Baseline | 0 | 0
  QTcF Interval >=60 msec Increase From Baseline | 0 | 0
  QTcF Interval 30-<60 msec Decrease From Baseline | 1 | 0
  QTcF Interval >=60 msec Decrease From Baseline | 0 | 0

6. Primary Outcome: Number of Participants With Confirmed Positive Anti-Drug Antibodies (ADAs)
Description: Assays for the determination of a positive immune response was performed. An antibody immune response was defined as a confirmed post-treatment positive enzyme-linked immunosorbent assay (ELISA) result in combination with a negative baseline sample ELISA result. ADA positive was defined as ADA titer (ie, the reciprocal of the highest dilution that gives a value equivalent to the cut point of the assay) >=4.32.
Time Frame: Baseline, and Days 15, 29, 57, 85 and Day 127/Early Termination
Population: The safety analysis population consists of all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 1 | 3
participants | 0 | 3

7. Secondary Outcome: Concentration of PF-06342674
Time Frame: Baseline through Day 127/Early Termination
Population: Participants in the placebo arm did not receive PF-06342674. Due to the early termination of the study, the small enrollment number and minimal data, concentration data were listed but not summarized, and pharmacokinetic (PK) parameters were not calculated for the PF-06342674 0.25 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Placebo | PF-06342674 0.25 mg/kg
Number analyzed (Participants) | 0 | 3
nanogram/milliliter (ng/ml) |  | NA (NA) — Due to the early termination of the study, the small enrollment number and minimal data, concentration data were not summarized.

ADVERSE EVENTS:
Time Frame: Baseline through Day 127/Early Termination.
Groups:
- PF-06342674: Participants received PF-06342674 0.25 mg/kg SC every other week during an 85-day treatment period.
Arm/Group | Placebo | PF-06342674
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1) | PF-06342674 (N=3)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the small enrollment number and minimal data, no statistical analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days.

Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.